CLINICAL TRIAL: NCT04994847
Title: APOE in the Predisposition to, Protection From, and Prevention of Alzheimer's Disease
Status: Enrolling by invitation | Type: Observational
Sponsor: Banner Health (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: NIH-APOE-R01-001
Record Dates: First submitted 2021-06-21; First posted 2021-08-06 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Amyloid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood will be collected annually and CSF collected every two years.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- APOE Unimpaired Observational Trial: 300 participants who are cognitively unimpaired; Yearly procedures: blood draw Every Two Year Procedures: cognitive and clinical assessments, CSF collection, MRI, and Tau and Amyloid PET scans
  Interventions: Drug: Amyloid and Tau PET

INTERVENTIONS:
Drug: Amyloid and Tau PET — NAV4694 and MK6240 PET scans completed every two years

SUMMARY:
The purpose of this study is to track changes in the brain related to Alzheimer's disease. The results from this study will be used to develop new approaches to prevent or delay the onset of memory and thinking problems associated with Alzheimer's.

DETAILED DESCRIPTION:
This study aims to establish, use, and extensively share a comprehensive longitudinal resource of genetic, non-genetic, and cognitive data, brain imaging and fluid biomarker measurements of amyloid-β, tau pathophysiology, neurodegeneration, and inflammation and biological samples to advance the study of cognitively unimpaired older adults at six levels of genetic risk for Alzheimer's disease due to their APOE genotype including understudied APOE2 and APOE4 homozygotes (HMs) at the lowest and highest risk and those APOE4 HMs and heterozygotes (HTs) who remain unimpaired at older ages due to unknown protective factors and spared pathophysiological effects despite their genetic risk.

Each participant will provide blood samples for clinical lab analysis, DNA, RNA, plasma, serum, and peripheral blood mononuclear cells (PBMCs) every 12 months; amyloid and tau PET scans, a nearly one hour battery of MRIs, a lumbar puncture (LP) for the collection of CSF samples, and a comprehensive battery of cognitive, behavioral, risk factor, and other assessments every 24 months. Extracted DNA will be used to characterize the participant's APOE genotype, screen for rare APOE variants that might make them eligible for other studies, and perform whole genome sequencing (WGS) and genome-wide genotyping.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 50 to 90 years old in good general health with no diseases expected to interfere with the study.
* Willing to undergo health and cognitive assessments, brain imaging sessions (MRI and PET), and collection and banking of blood with venipuncture and CSF by lumbar puncture for genetic research, biomarker research, and DNA banking.
* Determined to be cognitively unimpaired by PI (mechanisms may include verbal interview, participant or study partner reports or specific scores on cognitive assessments)

Exclusion Criteria:

* Participants with significant health issues or medical diseases that may interfere with participation, including infectious diseases that pose a risk to study personnel.
* For PET or MRI: Female participant who is pregnant, lactating, or of childbearing potential without a negative pregnancy test or being two years postmenopausal or surgically sterile.
* For MRI: Any contraindication for MRI including, but not limited to, pacemaker, aneurysm clips, artificial heart valves, ear implants, metal fragments or foreign objects in the eyes, skin, or body.
* For CSF collection: Medical or surgical contraindication for lumbar puncture (e.g. on anti-coagulant therapy or had prior lumbar spinal surgery).

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: For the Arizona APOE Cohort, we will establish a new longitudinal cohort of 300 cognitively unimpaired males and non-pregnant females, 50-90 years of age at the time of enrollment who will be enrolled based on their APOE genotype, age, other eligibility criteria, consent to participate in virtually all study procedures, and consent to provide a shared resource of anonymized data and biological samples for the research community. Participants will include 50 individuals with each of the six common APOE genotypes (known as 2/2, 2/3, 3/3, 2/4, 3/4, and 4/4) who are matched by age decile, sex, and educational level. Participants will not receive information about their APOE genotype from this project97 and will be studied under the auspicious of a single Institutional Review Board (IRB).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Amyloid PET Scan | 5 years
  The study will acquire NAV4694, a radiotracer specific to amyloid, PET scans to monitor total amyloid levels in the brain.
Tau PET Scan | 5 years
  The study will acquire MK6240, a radiotracer specific to Tau, PET scans to monitor total tau levels in the brain.
MRI | 5 years
  The study will acquire 3T MRI to look at brain volume

CONTACTS AND LOCATIONS:
Locations (1):
- Banner Alzheimer's Institute, Phoenix, Arizona, United States